CLINICAL TRIAL: NCT02933203
Title: Genetic Biomarkers of Executive Stress
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natalie Rasgon, Dr., Stanford University
Other Study IDs: 35668
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva or blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to examine whether stress predicts telomere length in individuals who hold executive-level positions. Telomeres are the caps at the end of each strand of DNA that may affect how cells age. Subjects will complete an online survey/interview and provide one blood sample or saliva samples. The goal is to understand whether stress predicts genetic markers of longevity.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the relationship between overall levels of stress and telomere length. It is hypothesized that the high stress group (based on the Perceived Stress Scale)compared to low stress group will have shorter telomere length. A secondary aim is to evaluate whether different types of stress have differing degrees of association with telomere length. An exploratory aim is to assess for gender differences in the association between stress and telomere length. The investigators are collecting a number of other measures, including demographics, work sector, perceived social support, and medical history, in order to adjust for potential confounders in the analysis.

This study is an extension of earlier work Dr. Rasgon has done with Dr. Elizabeth Blackburn at UCSF on the relationship between telomere length and mood outcomes. The investigators hope this study will add to the growing body of literature on stress and genetic markers of longevity, specifically how stress level and type is associated with telomere length. The increased understanding gained through this study may provide leads for predicting age-related diseases and early mortality in adults, thus benefiting others in the future.

ELIGIBILITY:
Inclusion Criteria:

1. People of either gender >18 years of age.
2. Subject hold executive-level position as defined as meeting the following criteria: having managerial responsibility over an organization or substantial part of an organization and/or having strategic influence over the direction of the organization
3. Subject or representative is willing to sign the consent for prior to enrollment into the study, and to participate in all aspects of the study. Prospective subject must give verbal assent if unable to sign written consent.
4. Adequate visual acuity to complete questionnaires.

Exclusion Criteria:

1. Subjects will be excluded if they have any of the following medical conditions:

   1. active heart disease
   2. acute psychiatric disorder (hospitalized in the past year)
   3. any medical condition deemed exclusionary by the Principal Investigator (PI)
2. Subject has a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within one year prior to screening.
3. Subject is currently taking any medication deemed exclusionary by PI.
4. Subject is pregnant, lactating, or planning to become pregnant during the study period.
5. Subject is participating or has participated in another research study within 30 days prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 subjects - individuals who hold executive-level positions. Participants are males and females, 18 or older, may be of any ethnic background. The investigators aim to recruit a diverse sample, reflective of the broader population.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Telomere Length | 1 day
  Subjects will come in for 1 visit to give a saliva or blood sample which will be used to measure telomere length.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Rasgon, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No